CLINICAL TRIAL: NCT01304030
Title: Improving Empathy and Relational Skills in Resident Physicians: A Randomized Controlled Trial
Brief Title: Improving Empathy and Relational Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Helen Riess, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 2009P001599; P001599 (Other Grant/Funding Number: Risk Management Foundation)
Record Dates: First submitted 2011-02-19; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Empathy
Keywords: Empathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): The experimental group receives Empathy Training. The control Group receives residency training as usual
  Interventions: Behavioral: Empathy Training Modules
- Control Group (Active Comparator): The control group receives residency training as usual
  Interventions: Behavioral: Residency Training as usual

INTERVENTIONS:
Behavioral: Empathy Training Modules — The Empathy Training Modules utilize translational research in emotion expression basic science, physiology of emotions, decoding facial expressions and self-regulation skills as pertaining to management of medical and surgical patients.
  Other Names: E.M.P.A.T.H.Y. (TM)
  Arms: Experimental Group
Behavioral: Residency Training as usual — Residents will receive their typical didactic and clinical education
  Other Names: Residency Training
  Arms: Control Group

SUMMARY:
Our research hypothesis is that residents who participate in the empathy and relational skills training modules will significantly improve in these skills as compared to a control group of residents who receive residency training as usual that includes the current standard training in the doctor-patient relationship. To evaluate this hypothesis, we will use a two-pronged approach to assessment. The first prong is the residents' self assessment of empathy and the second is from the patients' perspective.

DETAILED DESCRIPTION:
The study design is a randomized controlled trial assigning resident physicians (N=100) to either: (a) empathy and relational skills training; or (b) control group receiving standard residency training as usual. Over the course of six weeks, each resident physician in the experimental group will receive three 60-minute training sessions focused on empathy and relational skills (the residents assigned to the control condition will receive standard residency training as usual). The emerging neuroscience of emotions and empathy has provided the neurobiological and physiological bases for our Empathy Training Modules to enhance patient-doctor communication. These innovative modules provide the basic science and video modeling for empathy training. Based on cutting edge mirror neuron research, our training modules offer a novel approach to empathy and relational skills training that teaches physicians about the neurobiology and physiology of emotions in difficult or stressful patient interactions. We have developed professionally produced high definition training modules that portray difficult patient-physician interactions. Importantly, these videos also include physiological displays of emotion for both members of the dyad so that one can easily observe the degree to which patient and physician are physiologically concordant or discordant with one another. The empathy training is conducted at a deeper level of physiological awareness and regulation that promises to be more effective than traditional didactic teaching by integrating the technology of psychophysiology. The goal of raising awareness of physiologic indices during a patient-doctor interaction is to present an objective measure of emotional response to both explicit and implicit stimuli, which promises to be a powerful teaching tool to enhance empathic physician behaviors.

ELIGIBILITY:
Inclusion Criteria:

All medical and surgical residents who are based at Massachusetts General Hospital will be eligible to participate in the study.

Exclusion Criteria:

Residents who are rotating at sites other then Massachusetts General Hospital Residents who are on rotations that do not include clinical care

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Consultation and Relational Empathy Measure (CARE) measure | Up to 5 weeks (this is an average)
  At baseline: (1) Residents will complete the CARE measure (2) 10 patients in each resident's clinic will rate their encounter using the CARE Measure; (3) Residents will receive the Empathy and Relational Training Modules or residency training as usual. At the six-week endpoint: (4) residents will complete the CARE measure and (5) patients will complete the CARE measure after the clinic visit.

SECONDARY OUTCOMES:
Jefferson Empathy Scale Mehrabian Balanced Emotional Empathy Scale (BEES) (30 items) 2.Jefferson Empathy Scale (20 items 3. Neuroscience of Emotions Assessment 4. Ekman Facial Expression Decoding Assessment | Prospective
  The Mehrabian BEES Measures baseline empathy. The Jefferson Scale measures physician attitudes about the importance of empathy in clinical medical care. The Neuroscience of Emotions Test measures knowledge of basic science of emotions. The Ekman test measures ability to decode subtle facial expressions.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Riess, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Riess H. Empathy in medicine--a neurobiological perspective. JAMA. 2010 Oct 13;304(14):1604-5. doi: 10.1001/jama.2010.1455. No abstract available. PMID 20940387
- [Background] Riess H, Kelley JM, Bailey R, Konowitz PM, Gray ST. Improving empathy and relational skills in otolaryngology residents: a pilot study. Otolaryngol Head Neck Surg. 2011 Jan;144(1):120-2. doi: 10.1177/0194599810390897. PMID 21493400